CLINICAL TRIAL: NCT01284582
Title: Safety, Immunogenicity and Dose Response of ATH03, a New Vaccine Against the Cholesterol Ester Transfer Protein (CETP), in Healthy Male Subjects With High Density Lipoprotein Cholesterol (HDLc) Blood Concentrations Equal or Below 80 mg/dl
Brief Title: Safety, Immunogenicity and Dose Response of ATH03, a New Vaccine Against the Cholesterol Ester Transfer Protein (CETP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Affiris AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFF007
Record Dates: First submitted 2011-01-25; First posted 2011-01-27 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: HDL; Drug Safety
Keywords: CETP; Vaccine; Cholesterol; Inhibition
MeSH Terms: conditions — Inhibition, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ATH03 Group A (Experimental): ATH03, 10 µg, 0.2% Alum
  Interventions: Biological: ATH03
- ATH03 Group B (Experimental): ATH03, 30 µg, 0.2% Alum
  Interventions: Biological: ATH03
- ATH03 Group C (Experimental): ATH03, 100 µg, 0.2% Alum
  Interventions: Biological: ATH03

INTERVENTIONS:
Biological: ATH03 — 4 vaccinations

SUMMARY:
Phase 1 Study :Safety, Immunogenicity and Dose response of ATH03, a new vaccine against the cholesterol ester transfer protein (CETP), in healthy male subjects with high density lipoprotein cholesterol (HDLc) blood concentrations equal or below 80 mg/dl.

DETAILED DESCRIPTION:
This open-label Phase 1 study will be conducted in three groups of 12 subjects with HDLc blood concentrations equal or below 80 mg/dl at a single study center. 36 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* High density lipoprotein cholesterol (HDLc) blood concentrations equal or below 80 mg/dl

Exclusion Criteria:

* Clinically relevant pathological findings

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 264 days

SECONDARY OUTCOMES:
Immunogenicity | 264 days
Response to the various applied doses of ATH03 | 264 days

CONTACTS AND LOCATIONS:
Overall Officials: Achim Schneeberger, MD, Study Director — Affiris AG
Locations (1):
- Department for Clinical Pharmacology Medical University Vienna, Vienna, Vienna, Austria